CLINICAL TRIAL: NCT00383396
Title: Efficacy of Topical Cyclosporine 0.05% in the Prevention of Ocular Surface Inflammation Secondary to Pterygia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 1963
Record Dates: First submitted 2006-09-29; First posted 2006-10-03 (Estimated); Last update posted 2007-02-13 (Estimated); Status verified 2007-02

CONDITIONS: Pterygia
MeSH Terms: conditions — Pterygium | interventions — Cyclosporine

INTERVENTIONS:
Drug: Topical Cyclosporine

SUMMARY:
To Determine if topical cyclosporine 0.05% BID prevents recurrent inflammation and improves comfort in eyes with pterygia.

ELIGIBILITY:
Inclusion Criteria:

* pts with symptomatic pterygia unresponsive to palliative treatment.

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Barry Schechter, MD, Principal Investigator — Florida Eye Microsurgical Institute
Locations (1):
- Dr. Schechter, Boynton Beach, Florida, United States